CLINICAL TRIAL: NCT01756794
Title: Validation of an Accelerated Procedure of Selection in Early Liver Transplantation for Severe Alcoholic Hepatitis Not Responding to Medical Treatment QuickTransHAA.
Brief Title: Validation of the Procedure of Early Liver Transplantation in Alcoholic Hepatitis Resisting to Medical Treatment
Acronym: QuickTrans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-26; 2012-A00088-35 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2020-03

CONDITIONS: Alcoholic Hepatitis; Alcoholic Cirrhosis
Keywords: Alcoholic hepatitis; Liver transplantation; Alcohol relapse; Alcoholic cirrhosis
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Cirrhosis, Alcoholic | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transplantation of alcoholic hepatitis (Other): Patients of this arm will be selected for early liver transplantation for severe alcoholic hepatitis not responding to medical therapy. Selection process will be based on a specific algorithm and follow-up time will be 2 years
  Interventions: Procedure: Liver transplantation
- Transplantation for alcoholic cirrhosis (Other): Patients of this arm will be selected for liver transplantation for alcoholic cirrhosis using an abstinence period of 6 months. Outcome of these patients will be compared to that of patients transplanted for severe alcoholic hepatitis.
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation

SUMMARY:
The purpose of this study is to validate a strategy of identification of patients for early liver transplantation in severe alcoholic hepatitis. In this setting, short-term survival is very low (approx. 25% at 6 months) and a pilot study has suggested (mathurin et al. N Engl J Med 2011) that liver transplantation may be an option in very carefully selected patients who did not respond to medical treatment. This selection process deserves to be confirmed in a population of greater size. We hypothesized that patients selected with this process would have a same alcohol relapse rate after liver transplantation than patients transplanted for alcoholic cirrhosis and selected using a 6-month sobriety period

DETAILED DESCRIPTION:
Non-inferiority of alcohol relapse in early liver transplantation for severe alcoholic hepatitis as compared to patients transplanted for alcoholic cirrhosis.

ELIGIBILITY:
Inclusion Criteria (Group A):

* Age > 18 years
* Maddrey score > 32
* Liver biopsy confirming the diagnosis of alcoholic hepatitis
* Non-response to medical treatment: Lille score ≥ 0.45 at day 7, or early worsening of liver function (MELD score > 25) despite a low Lille score (< 0.45)
* Hospitalization stay < 1 month
* Algorithm score ≥ 220/250.

Inclusion Criteria (Group B):

* Age >18 years
* Diagnosis of alcoholic cirrhosis
* Alcoholic withdrawal of 6 months minimum before inscription on the transplant list
* MELD score ≥ 15 for patients with hepatocellular carcinoma responding to Milan criteria (1 node < 5 cm or 3 nodes < 3 cm)
* MELD score ≥ 20 preferably for patients not displaying hepatocellular carcinoma and that did not obtain an "expert" component
* No recommendation of MELD score for patients having obtained an "expert" component

Non-inclusion Criteria (Group A and B):

* Bacterial or viral infection uncontrolled by medical treatment
* Fungal or aspergillosis uncontrolled infection
* Hepatocellular carcinoma or invasive cancer
* Positive test for HBsAg, Positive test for HIV,Positive PCR for HCV
* Portal thrombosis
* Pregnancy or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of alcohol relapse in early liver transplantation for severe alcoholic hepatitis as compared to patients transplanted for alcoholic cirrhosis. | 2 years
  Aim is to demonstrate that alcohol relapse within the 2-year follow-up period in patients selected for early liver transplantation for severe alcoholic hepatitis is not inferior to that of patients transplanted for alcoholic cirrhosis using the 6-month sobriety period.

SECONDARY OUTCOMES:
Validation of the survival benefit of transplanted patients as compared to non-transplanted patients with severe alcoholic hepatitis | 2 years
  First secondary aim is to confirm the survival benefit of patients transplanted for severe alcoholic hepatitis as compared to patients suffering for severe alcoholic hepatitis not responding to medical treatment and not selected for early liver transplantation
Reproducibility of an algorithm of selection for candidates to liver transplantation | 2 years
  Second secondary aim is to evaluate the reproducibility of the algorithm for selection of candidates for liver transplantation in three centers
Incidence of alcohol relapse | 2 years
  Third secondary endpoint is to compare the incidence of alcohol relapse in patients selected for early transplantation for severe alcoholic hepatitis as compared to patients transplanted for alcoholic cirrhosis using the 6-month sobriety period rule
Pattern of alcohol relapse in the two groups of transplanted patients | 2 years
  Fourth secondary endpoint is to assess the pattern of alcohol relapse in the group of patients transplanted for severe alcoholic hepatitis to the group of patients transplanted for alcoholic cirrhosis using the 6-month sobriety rule.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Mathurin, MD,PhD, Study Chair — University hospital of Lille,
Locations (32):
- Belgium (4):
  - UZA, Antwerp, Edegem
  - ULB, Erasme, Brussels
  - Ghent
  - Hospital Sart Tilman, Liège
- France (28):
  - Univesity hospital, Amiens
  - University hospital, Angers
  - University hospital, Besançon
  - Hôpital Jean Verdier (AH-HP), Bondy
  - University hospital, Brest
  - University hospital, Caen
  - Univesity hospital, Chambray-lès-Tours
  - Hospital Antoine Béclère (Assistance Publique des Hôpiaux de Paris), Clamart
  - Hôpital Beaujon (AH-HP), Clichy
  - Hôpital Henri Mondor (AP-HP), Créteil
  - University hospital, Dijon
  - University hospital, Grenoble
  - University hospital, Lille
  - University hospital, Lyon
  - University Hospital, Montpellier
  - University hospital, Nancy
  - University hospital, Nantes
  - University hospital, Nice
  - Hôpital Saint Antoine (AP-HP), Paris
  - Hôpital de la Pitié-Salpétrière (AP-HP), Paris
  - Hôpital Cochin (AH-HP), Paris
  - University Hospital, Pessac
  - University hospital, Poitiers
  - University hospital, Reims
  - University hospital, Rennes
  - University Hospital, Strasbourg
  - University hospital, Toulouse
  - Hôpital Paul Brousse (AH-HP), Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Louvet A, Labreuche J, Moreno C, Vanlemmens C, Moirand R, Feray C, Dumortier J, Pageaux GP, Bureau C, Chermak F, Duvoux C, Thabut D, Leroy V, Carbonell N, Rolland B, Salame E, Anty R, Gournay J, Delwaide J, Silvain C, Lucidi V, Lassailly G, Dharancy S, Nguyen-Khac E, Samuel D, Duhamel A, Mathurin P; QuickTrans trial study group. Early liver transplantation for severe alcohol-related hepatitis not responding to medical treatment: a prospective controlled study. Lancet Gastroenterol Hepatol. 2022 May;7(5):416-425. doi: 10.1016/S2468-1253(21)00430-1. Epub 2022 Feb 23. PMID 35202597